CLINICAL TRIAL: NCT03776292
Title: Cardiopulmonary Effects of Prolonged Surgical Abdominal Retractors Application in Supine Versus Lateral Position During General Anesthesia
Brief Title: Cardiopulmonary Changes Prolonged Surgical Abdominal Retractors Application in Supine Versus Lateral Position
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abd Latif Ghanim, Associate Professor os anesthesia ICU & Pain medicine., Mansoura University
Other Study IDs: R.18.11.337
Record Dates: First submitted 2018-12-09; First posted 2018-12-14 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Cardio-pulmonary
Keywords: cardiac, output, pulmonary, compliance, bladder, Retractor.
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- supine position group= Group (S): 1st group of 20 patients will undergo urinary bladder cystectomy and orthotopic urinary diversion lying supine with ring abdominal retractors
  Interventions: Other: monitoring
- lateral position group = Group (L): 2nd group of 20 patients will undergo surgical open nephrectomy lying lateral position with self retaining abdominal retractors
  Interventions: Other: monitoring

INTERVENTIONS:
Other: monitoring — Primary outcome; composite 1ry outcome [1-Dynamic pulmonary compliance monitoring.2- Cardiac Index monitoring] during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups. Secondary outcome: Static lung compliance, Cardiac output, Stroke volume SV - stroke volume variability (SVV)-Cardiac performance index, O2 delivery DIO2. Noninvasive Intraoperative hemodynamic (MBP, HR, O2 saturation)] during and after surgical ring retractor application compared to the same variable reading prior retractor application and in between both groups.

SUMMARY:
Introduction: Dynamic and static compliance should be calculated as a routine part of ventilator monitoring. Dynamic and static compliance are 60-100 mL/cm H2O. A decrease in dynamic compliance without a change in the static compliance suggests an acute increase in airway resistance and can be assessed further by comparing peak pressure and plateau pressure. The normal gradient is approximately 10 cm H2O. A gradient >10 cm H2O may be secondary to endotracheal tube obstruction, mucous plugging, or bronchospasm. If volume is constant, acute changes in both dynamic and static compliance suggest a decrease in respiratory system compliance that may be caused by worsening increasing abdominal pressures. When static compliance is <25 mL/cm H2O, ventilator weaning may be difficult secondary to tachypnea during spontaneous breathing trials. (1) Aim of the work: to detect the cardiopulmonary burden of surgical ring retractors application during abdominal surgeries in supine versus lateral position (cancer bladder for supine position and open surgical nephrectomy for lateral position). Hypothesis: Abdominal retractors application would produce more cardiopulmonary instability during lateral position than during supine position for abdominal surgery. Patient & Methods: This comparative prospective randomized study, will be done on ASA I-II patients, both sexes, Age 18 - 65 year, to compare pulmonary compliance and cardiac performance before, during and after surgical self-retaining abdominal retractors application patients will be divided into 2 groups; 1st group (S) will undergo orthotropic cancer bladder diversion and the 2nd group (L) both supine and lateral position for open surgical nephrectomy for lateral position.

DETAILED DESCRIPTION:
Introduction: Dynamic and static compliance should be calculated as a routine part of ventilator monitoring. Dynamic and static compliance are 60-100 mL/cm H2O. A decrease in dynamic compliance without a change in the static compliance suggests an acute increase in airway resistance and can be assessed further by comparing peak pressure and plateau pressure. The normal gradient is approximately 10 cm H2O. A gradient >10 cm H2O may be secondary to endotracheal tube obstruction, mucous plugging, or bronchospasm. If volume is constant, acute changes in both dynamic and static compliance suggest a decrease in respiratory system compliance that may be caused by worsening increasing abdominal pressures. When static compliance is <25 mL/cm H2O, ventilator weaning may be difficult secondary to tachypnea during spontaneous breathing trials. (1) Aim of the work: to detect the cardiopulmonary burden of surgical ring retractors application during abdominal surgeries in supine versus lateral position (cancer bladder for supine position and open surgical nephrectomy for lateral position). Hypothesis: Abdominal retractors application would produce more cardiopulmonary instability during lateral position than during supine position for abdominal surgery. Patient & Methods: This comparative prospective randomized study, will be done on ASA I-II patients, both sexes, Age 18 - 65 year, to compare pulmonary compliance and cardiac performance before, during and after surgical self-retaining abdominal retractors application patients will be divided into 2 groups; 1st group (S) will undergo orthotropic cancer bladder diversion and the 2nd group (L) both supine and lateral position for open surgical nephrectomy for lateral position. Study will be done at Mansoura University Hospital, during the year 2018, for 4 month duration, starting predected date=1-11-2018 actual study start date=15-12-2018[ NB. by mistake in the 1st registration i have regestered the study protocol predicted time of study start but actually the study started on 15-12-2018 thats why i changed the date more than one time ] till 30-3-2019 after approval of IRB (Institutional Review Board), Mansoura Faculty of Medicine. Primary outcome; composite 1ry outcome [1-Dynamic pulmonary compliance.2- Cardiac Index] during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups. Secondary outcome: Static lung compliance, Cardiac output, Stroke volume SV - stroke volume variability (SVV)-Cardiac performance index CPI, O2 delivery DIO2. Noninvasive Intraoperative hemodynamic (MBP, HR, O2 saturation)] during and after surgical ring retractor application compared to the same variable reading prior retractor application and in between both groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* both sexes
* Age 18 - 65 year
* surgical time ≥ 6hours for Orthotopic urinary bladder diversion surgery for cancer bladder patients and 3 hours for open surgical nephrectomy.

Exclusion Criteria:

* Body mass index (BMI) greater than 35 kg. m-2.
* Asthma requiring bronchodilator therapy.
* Chronic Obstructive Pulmonary Disease, GOLD classification III and IV.
* Severe pulmonary disease.
* Hemodynamic instability (hypotension or tachycardia).
* History of congestive heart failure or New York Heart Association (NYHA) functional class IV
* Right ventricular dysfunction.
* Severe valvular heart disease.
* Intra-cardiac shunts.
* Intracranial hypertension.
* Cardiac rhythm other than regular sinus.
* Severe chronic kidney disease (glomerular filtration rate < 30 ml. min-1. 1.73 m2).
* Liver cirrhosis (Child Pugh class B or C).
* Pregnancy.
* Previous thoracic surgery (lobectomy, bilobectomy, or pneumonectomy).
* Lung metastatic surgery.
* Previous receiving chemotherapy.
* Emergency surgery.
* Preoperative need for invasive mechanical ventilation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -Patients admitted to the Urology Department, Mansoura Urology and Nephrology center, Faculty of medicine Mansoura University .
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
-non invasive Dynamic pulmonary compliance . | mean dynamic compliance at minutes 30,60,90,120,180,210 240 post retractor application compared to mean dynamic compliance at minutes 10,20,30,post endotracheal intubation(Basal Value preretractor application)
  dynamic pulmonary compliance during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups
Non invasive Cardiac Index | mean Non invasive Cardiac Index at minutes 30,60,90,120,180,210 240 post retractor application compared to mean Non invasive Cardiac Index at minutes 10,20,30,post endotracheal intubation(Basal Value preretractor application)
  Cardiac index monitoring during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups

SECONDARY OUTCOMES:
Static lung compliance | After endotracheal intubation recorded 3 times every 10 minutes -After Abdominal retractors application recorded every 30 minutes for 6 readings -After retractor removal 3 times every 10 minutes
  Static lung compliance during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups
Cardiac output. | After endotracheal intubation recorded 3 times every 10 minutes -After Abdominal retractors application recorded every 30 minutes for 6 readings -After retractor removal 3 times every 10 minutes
  Cardiac output. during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups
Stroke volume SV | After endotracheal intubation recorded 3 times every 10 minutes -After Abdominal retractors application recorded every 30 minutes for 6 readings -After retractor removal 3 times every 10 minutes
  Stroke volume SV. during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups
- stroke volume variability (SVV) | After endotracheal intubation recorded 3 times every 10 minutes -After Abdominal retractors application recorded every 30 minutes for 6 readings -After retractor removal 3 times every 10 minutes
  Stroke volume variability (SVV)during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups
-Cardiac performance index CPI | After endotracheal intubation recorded 3 times every 10 minutes -After Abdominal retractors application recorded every 30 minutes for 6 readings -After retractor removal 3 times every 10 minutes
  Cardiac performance index during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups
Oxygen delivery DIO2 | After endotracheal intubation recorded 3 times every 10 minutes -After Abdominal retractors application recorded every 30 minutes for 6 readings -After retractor removal 3 times every 10 minutes
  Oxygen delivery DIO2 during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups
. Noninvasive Intraoperative MBP | After endotracheal intubation recorded 3 times every 10 minutes -After Abdominal retractors application recorded every 30 minutes for 6 readings -After retractor removal 3 times every 10 minutes
  Noninvasive Intraoperative MBP during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups
HR | After endotracheal intubation recorded 3 times every 10 minutes -After Abdominal retractors application recorded every 30 minutes for 6 readings -After retractor removal 3 times every 10 minutes
  HR during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups
arterial O2 saturation(SaO2%) | After endotracheal intubation recorded 3 times every 10 minutes -After Abdominal retractors application recorded every 30 minutes for 6 readings -After retractor removal 3 times every 10 minutes
  SaO2 saturation during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups
End tidal Co2 EtCO2 | After endotracheal intubation recorded 3 times every 10 minutes -After Abdominal retractors application recorded every 30 minutes for 6 readings -After retractor removal 3 times every 10 minutes
  End tidal Co2 EtCO2 during and after surgical retractor application compared to the same variables reading prior retractor application and in between both groups

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Ghanem, A professor, Principal Investigator — Mansoura Univeristy
Locations (1):
- Mansoura faculty of Medicine- Mansoura Urology and nephrology center, Al Mansurah, Dakahlia Governorate, Egypt